CLINICAL TRIAL: NCT03757091
Title: Flexible Scope Intubation vs.Flexible Scope Intubation and Video Laryngoscopy Combination: A Prospective Randomized Clinical Trial
Brief Title: Flexible Intubation Scope With or Without Video Laryngoscope in Supporting Endotracheal Tube Placement in Patients With Head and Neck Cancer Before Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0661; NCI-2018-02698 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0661 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Laryngoscopy; Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (flexible intubation scope) (Active Comparator): Patients undergo flexible scope intubation up to 2 attempts following induction of general anesthesia and adequate manual ventilation. In case of failed 2 attempts, patients undergo a third attempt utilizing another technique or device.
  Interventions: Procedure: Tracheal Intubation
- Arm B (flexible intubation scope,video laryngoscope) (Experimental): Patients undergo flexible scope intubation and video laryngoscopy up to 2 attempts following induction of general anesthesia and adequate manual ventilation. In case of failed 2 attempts, patients undergo a third attempt utilizing another technique or device.
  Interventions: Device: Laryngoscopy; Procedure: Tracheal Intubation

INTERVENTIONS:
Device: Laryngoscopy — Undergo video laryngoscopy
  Arms: Arm B (flexible intubation scope,video laryngoscope)
Procedure: Tracheal Intubation — Undergo flexible scope intubation

SUMMARY:
This trial studies how well flexible intubation scope with or without video laryngoscope works in supporting endotracheal tube placement in patients with head and neck cancer before surgery. Flexible intubation scope and video laryngoscope are devices that have a small camera to help the doctor see the patient's airway on a screen. Both devices may help the doctor who gives anesthesia prevent complications from placing the breathing tube (such as pain or mouth injury).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the rates of difficult endotracheal tube (ETT) placement using a flexible intubation scope (FIS) versus a combination of flexible intubation and video laryngoscopy in difficult airway management.

SECONDARY OBJECTIVES:

I. To compare the ease of using a flexible intubation scope (FIS) with and without the use of the video laryngoscope (VL).

II. Total time for securing the airway.

III. Number of attempts required for intubation.

IV. Rate of failure at intubation.

V. Incidence of desaturation.

VI. Assessment for hoarseness, sore mouth, neck, or jaw, dysphonia, dysphagia, lip injury, tongue injury, or tooth damage.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo flexible scope intubation up to 2 attempts following induction of general anesthesia and adequate manual ventilation. In case of failed 2 attempts, patients undergo a third attempt utilizing another technique or device.

ARM B: Patients undergo flexible scope intubation and video laryngoscopy up to 2 attempts following induction of general anesthesia and adequate manual ventilation. In case of failed 2 attempts, patients undergo a third attempt utilizing another technique or device.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥ 18 years of age
* All surgical patients with known or suspected difficult airways that meet at least three (3) of the Difficult Airway criteria [Mallampati III-IV, Neck circumference > 40 cm, Sternomental distance < 12 cm, Thyromental distance < 6 cm, Mouth opening < 4 cm, BMI ≥ 35 kg/m2, Upper Lip Bite Test - ULBT (class III)] or history of radiation to the head and neck area or oral pathology obstructing the glottic view
* American Society of Anesthesiology (ASA) I-IV
* Has provided written informed consent

Exclusion Criteria:

* Active bleeding from nasopharynx or oropharynx
* Trismus
* Oral pathology obstructing the glottic view
* Planned awake or nasal intubation
* Neuromuscular Blockade (NMB) contraindicated post-induction
* Emergency endotracheal intubation and patients intubated pre and post-surgery
* Surgical procedures such as Tracheostomy, Laryngectomy, Esophagectomy
* Patient refusal or inability to consent for study participation
* American Society of Anesthesiology (ASA) V
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Carin Hagberg, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Main OR procedure daily schedule will be used for patient selection. Once eligibility of a study candidate has been identified, the study coordinator will be informed to start the patient interview and obtain written informed consent.
Groups:
- Flexible Intubation Scope (FIS): control group will utilize FIS (flexible intubation scope)
- Flexible Intubation Scope + Video Laryngoscope (FIS+VL): treatment group will utilize FIS+VL (flexible intubation scope + video laryngoscope)
Period: Overall Study
Arm/Group | Flexible Intubation Scope (FIS) | Flexible Intubation Scope + Video Laryngoscope (FIS+VL)
Started | 69 | 66
Completed | 64 | 58
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexible Intubation Scope (FIS) | Flexible Intubation Scope + Video Laryngoscope (FIS+VL) | Total
Number analyzed (Participants) | 69 | 66 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 41 | 77
  >=65 years | 33 | 25 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.20 (11.84) | 59.26 (13.97) | 61.23 (12.905)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 39 | 39 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 69 | 66 | 135

OUTCOME MEASURES:

1. Primary Outcome: Difficult Endotracheal Tube (ETT) Placement
Description: Defined as the number of participants with any of the following during initial intubation attempt.1 Intubation time exceeding 60 seconds, 2. Failure to intubate on the first attempt, 3. Provider assessment of intubation as difficult or unsuccessful.
Time Frame: intubation time, up to 3 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Flexible Intubation Scope (FIS) | Flexible Intubation Scope + Video Laryngoscope (FIS+VL)
Number analyzed (Participants) | 67 | 63
Participants
  Yes | 40 | 29
  No | 27 | 34

2. Secondary Outcome: Intubation Time
Description: Time from induction to successful intubation
Time Frame: time captured when FIS passed the lips to CO2 confirmation
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Flexible Intubation Scope (FIS) | Flexible Intubation Scope + Video Laryngoscope (FIS+VL)
Number analyzed (Participants) | 64 | 58
seconds | 58.37 [51.44 to 65.30] | 50.92 [44.04 to 57.80]

3. Secondary Outcome: Number of Intubation Attempts
Description: Number of Intubation Attempts
Time Frame: intubation time, up to 3 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Flexible Intubation Scope (FIS) | Flexible Intubation Scope + Video Laryngoscope (FIS+VL)
Number analyzed (Participants) | 64 | 58
Participants
  1 | 50 | 54
  2 or more | 14 | 4

4. Secondary Outcome: Rate of Failure at Intubation
Description: Failed Airway Rate
Time Frame: during intubation process/attempt
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flexible Intubation Scope (FIS) | Flexible Intubation Scope + Video Laryngoscope (FIS+VL)
Number analyzed (Participants) | 64 | 58
percentage of participants | 7.81 [7.76 to 26.86] | 1.72 [0.42 to 11.91]

5. Secondary Outcome: Ease of Intubation (Provider Assessment)
Description: The number of people who had 1= extremely easy, 2=somewhat easy, 3=resistance, 4= difficult, 5= unsuccessful (for both groups)
Time Frame: duration of intubation attempt
Measure: Count of Participants; unit: Participants
Arm/Group | Flexible Intubation Scope (FIS) | Flexible Intubation Scope + Video Laryngoscope (FIS+VL)
Number analyzed (Participants) | 67 | 64
Participants
  1= extremely easy | 31 | 40
  2=somewhat easy | 14 | 14
  3=resistance | 9 | 6
  4= difficult | 2 | 2
  5= unsuccessful | 11 | 2

ADVERSE EVENTS:
Time Frame: From induction to one hour after PACU arrival, up to 6 hours
Arm/Group | Flexible Intubation Scope (FIS) | Flexible Intubation Scope + Video Laryngoscope (FIS+VL)
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/66
Other Adverse Events (participants affected / at risk) | 0/69 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03757091/Prot_SAP_000.pdf